CLINICAL TRIAL: NCT00241553
Title: Efficacy of Esomeprazole 40 mg Once Daily Versus Placebo or Esomeprazole 20 mg Once Daily Versus Placebo in Prevention of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs Including COX-2 Selective NSAIDs
Brief Title: Esomeprazole for Prevention of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9617C00004; SH-NEN-0004
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: NSAIDs; Upper GI Symptoms
MeSH Terms: interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
This study was a multicentre, double-blind, randomised, placebo-controlled parallel group study consisting of 4 visits over a period of 6 months. The primary variable was to assess theefficacy of esomeprazole 40 mg orally qd (E40) or esomeprazole 20 mg orally qd (E20) versus placebo orally qd after 6 months of treatment for the prevention of relapse of upper GI symptoms associated with NSAID use, including COX-2 selective NSAIDs, in patients receiving daily NSAID therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Completed the SH-NEN-0003 study with relief of upper GI symptom. Relief is defined as "last 7 days with a diary assessment of None or Minimal, but allowing up to 2 days to be rated as Mild during the 7-day period".
* A clinical diagnosis of a chronic condition (e.g., osteoarthritis or rheumatoid arthritis) that requires continuous daily NSAID treatment for at least 6 months. Daily NSAID treatment is defined as taking the prescribed dose for at least 5 of 7 days in any given week and can include COX-2 selective NSAIDs, multiple NSAIDs, and high-dose NSAIDs.
* Daily NSAID treatment dose and type:
* Must have been stable for at least 9 weeks prior to inclusion
* Are expected to remain stable for the duration of the study.
* Must be administered orally. If more than one type of NSAID treatment is used, at least one type must be administered orally.
* Hp negative on Histology performed at baseline endoscopy in the study SHNEN-0003.

Exclusion Criteria:

* Discontinuation from study SH-NEN-0003
* Pain, discomfort or burning in the upper abdomen precipitated by exercise or relieved by defecation.
* Pain, discomfort or burning in the upper abdomen not associated with the use of NSAIDs, including COX-2 selective NSAIDs.
* Pregnancy or lactation. Women of childbearing potential must maintain effective contraception during the study period as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276
Dates: Start 2001-04; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of esomeprazole versus placebo through 6 months of treatment for the prevention of relapse of upper GI symptom associated with NSAID use

SECONDARY OUTCOMES:
To assess the safety & tolerability of esomeprazole versus placebo when administered for 6 months to patients receiving daily NSAID therapy.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (136):
- United States (31):
  - Research Site, Tallassee, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Garden Grove, California
  - Research Site, Orange, California
  - Research Site, Bradenton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Hollywood, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tavares, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Nampa, Idaho
  - Research Site, Elkhart, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Newburgh, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Hollywood, Maryland
  - Research Site, Butte, Montana
  - Research Site, Princeton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Endwell, New York
  - Research Site, Hewlett, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Jackson, Tennessee
  - Research Site, Waco, Texas
  - Research Site, Edmonds, Washington
  - Research Site, Olympia, Washington
  - Research Site, Greenfield, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Australia (8):
  - Research Site, Five Dock, New South Wales
  - Research Site, Various Cities, New South Wales
  - Research Site, Carina Heights, Queensland
  - Research Site, Kippa-Ring, Queensland
  - Research Site, Various Cities, South Australia
  - Research Site, Various Cities, Tasmania
  - Research Site, Ivanhoe, Victoria
  - Research Site, Various Cities, Victoria
- Canada (16):
  - Research Site, Edmonton, Alberta
  - Research Site, Quesnel, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sainte-Foy, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Czechia (4):
  - Research Site, Hlu¿ín
  - Research Site, Ostrava
  - Research Site, Ostrava - T¿ebovice
  - Research Site, Prague
- Italy (8):
  - Research Site, Bari, BA
  - Research Site, Genova, GE
  - Research Site, Milan, MI
  - Research Site, Vicenza, VI
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Verona
- Norway (12):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Bærum Postterminal
  - Research Site, Gjøvik
  - Research Site, Horten
  - Research Site, Lillehammer
  - Research Site, Nesttun
  - Research Site, Oslo
  - Research Site, Sandvika
  - Research Site, Skien
  - Research Site, Stavanger
  - Research Site, Tromsø
- Poland (5):
  - Research Site, Bia¿ystok
  - Research Site, Bydgoszcz
  - Research Site, Sopot
  - Research Site, Warsaw
  - Research Site, Wrze¿nia
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Pie¿¿any
- South Africa (3):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Johannesburg
- Sweden (17):
  - Research Site, Bredbyn
  - Research Site, Gävle
  - Research Site, Karlskrona
  - Research Site, Kungälv
  - Research Site, Lidköping
  - Research Site, Malmo
  - Research Site, Oskarshamn
  - Research Site, Örnsköldsvik
  - Research Site, Östersund
  - Research Site, Rättvik
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Trehörningsjö
  - Research Site, Trollhättan
  - Research Site, Varberg
  - Research Site, Värnamo
  - Research Site, Västervik
- United Kingdom (29):
  - Research Site, Reading, Berks
  - Research Site, Spennymoor, Co. Durham
  - Research Site, Woking, Surrey
  - Research Site, Trowbridge, Wiltshire
  - Research Site, Ashford
  - Research Site, Audley
  - Research Site, Bath
  - Research Site, Bradford Upon Avon
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Crawley
  - Research Site, Ely
  - Research Site, Folkestone
  - Research Site, Glasgow
  - Research Site, Kilmarnock
  - Research Site, Leigh
  - Research Site, Mansfield
  - Research Site, Nottingham
  - Research Site, Pontefract
  - Research Site, Royal Tunbridge Wells
  - Research Site, Shrewsbury
  - Research Site, Stafford
  - Research Site, Swansea
  - Research Site, Trowbridge
  - Research Site, Watford
  - Research Site, Wigston
  - Research Site, Woking
  - Research Site, Worsley
  - Research Site, Yoxall

REFERENCES:
- [Derived] Hawkey CJ, Talley NJ, Scheiman JM, Jones RH, Langstrom G, Naesdal J, Yeomans ND; NASA/SPACE author group. Maintenance treatment with esomeprazole following initial relief of non-steroidal anti-inflammatory drug-associated upper gastrointestinal symptoms: the NASA2 and SPACE2 studies. Arthritis Res Ther. 2007;9(1):R17. doi: 10.1186/ar2124. PMID 17391505